CLINICAL TRIAL: NCT05861609
Title: Pain Medication Tapering for Patients With Persistent Spinal Pain Syndrome Type 2, Treated With Spinal Cord Stimulation.
Acronym: PIANISSIMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moens Maarten (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, Principal Investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIANISSIMO
Record Dates: First submitted 2023-05-06; First posted 2023-05-17 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Persistent Spinal Pain Syndrome Type 2; Spinal Cord Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both the outcome assessors as well as the investigator (statistician) will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No pain medication tapering (usual care) (Active Comparator): Usual care
  Interventions: Procedure: Usual care
- Standardized pain medication tapering (Active Comparator): Standardized pain medication tapering
  Interventions: Procedure: Standardized pain medication tapering
- Personalized pain medication tapering (Active Comparator): Personalized pain medication tapering
  Interventions: Procedure: Personalized pain medication tapering

INTERVENTIONS:
Procedure: Usual care — Usual care with respect to Spinal Cord Stimulation implantation
  Arms: No pain medication tapering (usual care)
Procedure: Standardized pain medication tapering — A standardized pain medication tapering program before Spinal Cord Stimulator implantation.
  Arms: Standardized pain medication tapering
Procedure: Personalized pain medication tapering — A personalized pain medication tapering program before Spinal Cord Stimulator implantation.
  Arms: Personalized pain medication tapering

SUMMARY:
The primary objective of the study is to examine whether there is a difference in disability after 12 months of Spinal Cord Stimulation (SCS) in patients with Persistent Spinal Pain Syndrome Type 2 (PSPS T2) after receiving a standardized pain medication tapering protocol before SCS implantation, a personalized pain medication tapering protocol before SCS implantation, or no tapering protocol before SCS implantation. The secondary objective of the study is to examine whether there is a difference after 12 months of SCS in PSPS T2 patients after receiving a standardized pain medication tapering protocol before SCS implantation, a personalized pain medication tapering protocol before SCS implantation, or no tapering protocol before SCS implantation on pain intensity, health-related quality of life, participation, domains affected by substance use, anxiety and depression, medication use, psychological constructs, sleep, central sensitization, and healthcare expenditure.

DETAILED DESCRIPTION:
Persistent Spinal Pain Syndrome Type II (PSPS T2) is a condition in which patients are suffering from persistent low back pain, despite previously performed surgical interventions. One way to help patients to alleviate their pain, is with Spinal Cord Stimulation (SCS). SCS is able to provide pain relief and a decrease in disability but also to decrease the amount of pain medication and more specifically opioid intake. Nevertheless, the number of patients that can eventually totally omit the use of opioids is rather limited.

In this trial, we will investigate the effect of a pain medication tapering program before starting the SCS trajectory as the new treatment strategy for patients implanted with SCS. This allows us to tackle the high burden of patients that are taking a lot of pain medication by proceeding towards a more logical treatment plan for a costly and debilitating condition.

A three-arm multicenter randomized controlled trial will be conducted to evaluate whether there is a difference in disability (primary outcome) after 12 months of SCS in PSPS T2 patients after receiving a standardized pain medication tapering protocol before SCS implantation, a personalized pain medication tapering protocol before SCS implantation, or no tapering protocol before SCS implantation. Two different pain medication tapering programs (standardized versus personalized tapering) will be evaluated in this project. Pain medication tapering will be provided to 130 patients during a hospital stay, compared to 65 patients who do not undergo pain medication tapering before SCS implantation. Besides disability as primary outcome measure, several secondary outcome measurements will be collected namely pain intensity, health-related quality of life, participation, domains affected by substance use, anxiety and depression, medication use, psychological constructs, sleep, central sensitization and health expenditure. Outcome measurements will be collected at baseline, and after 1 month, 3, 6 and 12 months of SCS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PSPS T2, defined as patients suffering from neuropathic pain of radicular origin with pain in the lower back and/or leg(s), of an intensity of at least 4/10 on the Numeric Rating Scale, for a period of at least 6 months after a minimum of one anatomically successful spinal surgery and being refractory to conservative treatment (according to Belgian reimbursement rules from January 1st, 2018)
* Patients need to be scheduled for SCS to be eligible for participation in the study
* Currently taking opioids
* 18 years and older
* Speaking and reading Dutch or French

Exclusion Criteria:

* Being actively treated for cancer.
* Having a life expectancy below 6 months.
* Receiving intrathecal drug delivery.
* Patients with contraindications for Clonidine (e.g., known hypotension which requires medication) or for Buprenorphine/Naloxone (e.g., severe respiratory insufficiency, hepatic insufficiency).
* Epilepsy treated by Pregabalin.
* Currently using benzodiazepines at more than 40 mg diazepam-equivalents per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Disability | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation
  Disability, evaluated with the Oswestry Disability Index

SECONDARY OUTCOMES:
Pain intensity | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  Pain intensity will be evaluated using a Visual Analogue Scale (100 mm).
Health-related Quality of Life | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  Health-related quality of life will be assessed using the Euro Quality of Life with five dimensions and five levels.
Participation | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  The Impact on Participation and Autonomy Questionnaire is used to evaluate participation.
Drug related patient characteristics and problems | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  The Measurements in the Addictions for Triage and Evaluation is used assess drug related patient characteristics and problems.
Opioid craving | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  Opioid craving will be assessed with the Visual Analogue Scale for Opioid Craving.
Risk for aberrant medication-related behaviour | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  The Current Opioid Misuse Measure is used to evaluate the risk for aberrant medication-related behaviour.
Medication use | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  The Medication Quantification Scale III is used to quantify pain medication use.
Healthcare utilization | The change in healthcare utilization starting from the baseline screening up to 12 months after the intervention.
  Healthcare utilization is investigated by two means: expenditures associated with in-hospital care are inventoried using the hospital claims data whereas other costs are collected through self-reported (diaries and questionnaires).
Anxiety and depression | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  The Hospital Anxiety and Depression Scale is used to assess feelings of anxiety and depression.
General Self-Efficacy | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  Perceived self-efficacy is evaluated using the General Self-Efficacy Scale.
Pain Catastrophizing | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  With the Pain Catastrophizing Scale, catastrophizing thoughts or feelings accompanying the previously experienced pain are evaluated.
Coping | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  The Multidimensional Pain Inventory is used to assess the participants coping strategy profile.
Sleep quality | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  The Pittsburgh Sleep Quality Index is used to assess sleep quality.
Symptoms of Central Sensitization | The change between the baseline assessment and the evaluation 1 month, 3 months, 6 months, and 12 months after receiving Spinal Cord Stimulation.
  To assess symptoms associated with central sensitization, the Central Sensitization Inventory is used.

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Jette
  - Heilig Hart Ziekenhuis Lier, Lier
  - AZ Delta, Roeselare

REFERENCES:
- [Derived] Moens M, Crunelle CL, Putman K, Wuyts E, Bultinck F, Van Puyenbroeck H; PIANISSIMO consortium; Goudman L. Pain medication tapering for patients with Persistent Spinal Pain Syndrome Type II, treated with Spinal Cord Stimulation: A RCT-study protocol of the PIANISSIMO study. PLoS One. 2024 Aug 12;19(8):e0302842. doi: 10.1371/journal.pone.0302842. eCollection 2024. PMID 39133680